CLINICAL TRIAL: NCT06966687
Title: Protective Effect of Ulinastatin and Thymosin α1 Against Negative Immune Dysregulation and Organ Dysfunction After Acute Aortic Dissection Surgery (PANDA XI)
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Collaborators: Beijing Anzhen Hospital (Other); West China Hospital (Other); Shanghai East Hospital,Tongji University School of Medicine (Unknown); The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Hong Liu, Principal Investigator of Department of Cardiovascular Surgery, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PANDA XI
Record Dates: First submitted 2025-05-04; First posted 2025-05-13 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Aortic Dissection; Aortic Dissection Aneurysm
Keywords: Aortic Dissection; inflammation
MeSH Terms: conditions — Aortic Dissection; Inflammation | interventions — urinastatin

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UT Group (Experimental): Ulinastatin (100000U TID for 5 days) and Thymosin alpha 1 (1.6 mg q12h for 5 days) immediately after surgery
  Interventions: Drug: Ulinastatin and Thymosin α1
- Control Group (Active Comparator): Ulinastatin (100000U TID for 5 days) immediately after surgery
  Interventions: Drug: Ulinastatin only

INTERVENTIONS:
Drug: Ulinastatin and Thymosin α1 — Ulinastatin (100000U TID for 5 days) and Thymosin alpha 1 (1.6 mg q12h for 5 days) immediately after surgery
  Arms: UT Group
Drug: Ulinastatin only — Ulinastatin (100000U TID for 5 days) immediately after surgery
  Arms: Control Group

SUMMARY:
Systemic inflammatory response syndrome (SIRS) and multiple organ dysfunction syndrome (MODS) are the major causes of death in patients with acute aortic syndrome (AAS). Therefore, the prevention of SIRS and MODS is of great clinical value, and immunomodulatory therapy with thymosin alpha

1 in addition to antiinflammatory treatment may be beneficial. This study was designed to test the hypothesis that the administration of Ulinastatin and Thymosin α1 during the acute phase of AAS will result in a reduced incidence of SIRS and MODS.

ELIGIBILITY:
Inclusion Criteria:

* The patients are conformed to 2010 ACC/AHA guidelines for the diagnosis and treatment of thoracic aortic disease (TAD) within two weeks of onset;
* Patients with acute aortic syndrome confirmed clinically and radiologically and planning to undergo emergency surgery were enrolled.
* The patients' age between 18 ~90 years old.
* Agree to participate in the study and sign the informed consent.

Exclusion Criteria:

* Patients allergic to Thymosin α1 or Ulinastatin;
* Lactating women and pregnant women;
* Patients with mental diseases, drug and alcohol dependence;
* Refuse to participate in this study and refuse to sign the informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The mean Sequential Organ Failure Assessment (SOFA) score of 7 days after surgery | within the prior 7 days after surgery.
  The occurrence of new-onset organ failure and new-onset persistent organ failure (Sequential Organ Failure Assessment (SOFA) score. New-onset is defined as events that occur after randomization and not present 24 hours before randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Yong-feng Shao, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (4):
- China (4):
  - Beijing Anzhen Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Shanghai East Hospital Tongji University, Shanghai, Shanghai Municipality
  - West China Hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Liu D, Yu Z, Yin J, Chen Y, Zhang H, Xin F, Fu H, Wan B. Effect of ulinastatin combined with thymosin alpha1 on sepsis: A systematic review and meta-analysis of Chinese and Indian patients. J Crit Care. 2017 Jun;39:259-266. doi: 10.1016/j.jcrc.2016.12.013. Epub 2016 Dec 27. PMID 28069319